CLINICAL TRIAL: NCT05156658
Title: Pharmacokinetic Interactions of Etonogestrel (ENG) Subdermal Implants with Long-Acting (LA) Cabotegravir (CAB-LA) and LA Rilpivirine (RPV-LA) (CARLA) in Participants of Reproductive Potential
Brief Title: Pharmacokinetic Interactions of ENG Subdermal Implants with Long-Acting Cabotegravir (CAB-LA) and LA Rilpivirine (RPV-LA) (CARLA)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol's question was answered elsewhere and very low site interest in the trial
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5392; UM1AI068636 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — etonogestrel; Endoglin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: With HIV receiving Monthly CARLA: ENG subcutaneous implant (Active Comparator): Participants with HIV-1 receiving monthly cabotegravir-long acting and rilpivirine-long acting (CARLA) (not provided by the study) will receive ENG implant immediately after enrollment.
  Interventions: Drug: Etonogestrel (ENG) Subdermal Implants
- Group B: Without HIV: ENG subcutaneous implant (Active Comparator): Participants without HIV-1 will receive ENG implant immediately after enrollment.
  Interventions: Drug: Etonogestrel (ENG) Subdermal Implants

INTERVENTIONS:
Drug: Etonogestrel (ENG) Subdermal Implants — Etonogestrel is available as a single, white/off-white, soft, radiopaque, flexible, ethylene vinyl acetate copolymer implant, 4 cm in length and 2 mm in diameter containing 68 mg of etonogestrel. Store at 25°C (77°F); excursions permitted between 15 and 30°C (59-86°F) [see USP Controlled Room Temperature]. Avoid storing ENG at temperatures above 30°C (86°F).

SUMMARY:
The purpose of this pharmacokinetic (PK) trial is to evaluate whether the ENG implant, a long-acting birth control method, is tolerable and effective for adults with HIV who are taking long-acting cabotegravir (CAB-LA) and long-acting rilpivirine (RPV-LA). Access to safe and effective birth control for adults with HIV is important because it may result in fewer infants exposed to HIV in the womb or born with HIV. Researchers believe that people of childbearing potential need access to birth control options that do not need to be negotiated with a partner.

ELIGIBILITY:
Inclusion Criteria:

* Last menstrual period started ≤35 days prior to study entry. If the start of the last menstrual period was >35 days prior to study entry, and the individual has been using hormonal contraception for at least 30 days prior to study entry, individual is eligible. If the start of the last menstrual period was >35 days prior to study entry, and the individual has not been using hormonal contraception for at least 30 days prior to study entry, serum follicle-stimulating hormone (FSH) must be ≤40 mIU/mL.
* Negative serum or urine pregnancy test (urine test must have a sensitivity of ≤25 mIU/mL) within 48 hours prior to study entry by any US clinic or laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent, or is using a point-of-care (POC)/ CLIA-waived test, or at any network-approved non-US laboratory or clinic that operates in accordance with Good Clinical Laboratory Practice (GCLP) and participates in appropriate external quality assurance programs.
* Willingness and ability to have ENG implant placed per section 5.1.2.
* The following laboratory values obtained within 30 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that operates in accordance with GCLP and participates in appropriate external quality assurance programs.

  * Hemoglobin ≥8.0 g/dL
  * Creatinine clearance >60 mL/min/1.73m2

    o Refer to the calculator located on the Frontier Science website (at www.frontierscience.org): Calculated Creatinine Clearance - Cockcroft-Gault Equation (Adult).
  * Aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) <2.5 x upper limit of normal (ULN)
  * Alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) <2.5 x ULN
  * Total bilirubin <1.5 x ULN
  * Platelet count ≥50,000 platelets/mm3
* Ability and willingness of the individual to provide informed consent.
* HIV status, documented by one of the following, based on group:

Group A: Presence of HIV-1 Infection Documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

OR

Group B: Absence of HIV-1 infection Documented by any licensed rapid HIV test or HIV E/CIA test kit obtained within 30 days prior to study entry.

NOTE: The term "licensed" refers to a US FDA-approved kit or, for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally.

WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

* Body Mass Index (BMI) (kg/m2) available from weight/height measurements obtained within 30 days prior to study entry.

NOTE: Refer to the BMI Index calculator located on the Frontier Science website.

Group A-specific Additional Inclusion Criteria (Participants with HIV)

* Willingness to adhere to the following contraception requirements.

  a. Individuals who are participating in sexual activity that could lead to pregnancy must agree to use a non-hormonal method of contraception in addition to the ENG implant while participating in the study. Acceptable forms of contraception include:
  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Non-hormonal intrauterine device (IUD)
  * Bilateral tubal ligation
  * Male partner vasectomy
* Receiving monthly CARLA for ≥24 weeks immediately prior to study entry.

NOTE A: Oral CAB+RPV bridging that was used to cover one or more missed injection(s) is acceptable. If the individual missed an injection within the 24 weeks prior to study entry without oral bridging of CAB+RPV until the next injection was received, this would be defined as a missed dose and is exclusionary. The last dose of oral CAB+RPV must have occurred more than 4 weeks prior to study entry, with an intervening injection of CARLA since that oral dose.

NOTE B: For individuals co-enrolling from a study through which they are receiving CARLA, sites must document the study number and the participant's identifier on that study.

* No documentation of HIV-1 plasma RNA of ≥200 copies/mL obtained within 90 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that is VQA certified.
* HIV-1 plasma RNA of <200 copies/mL obtained within 30 days prior to study entry by any US laboratory that has a CLIA certification or its equivalent, or at any network-approved non-US laboratory that is VQA certified.
* Agreement not to change ART regimen (CARLA) for the duration of the study including the frequency of CARLA administration from monthly to every 8 weeks.

Exclusion Criteria:

* Hysterectomy or bilateral oophorectomy.
* Within 30 days postpartum at study entry.
* Currently breastfeeding or planning to become pregnant during the study.
* Participated in sexual activity that could lead to pregnancy in the 14 days prior to study entry without contraception, as reported by individual.
* Plans to use sex hormonal therapy, including but not limited to hormonal contraceptives, other than the ENG implant, during the study.
* The study puts the individual at unacceptable risk based on the judgment of the site investigator.
* Current or past history of thrombosis or thromboembolic disorder(s).
* Current or past history of breast, liver, or cervical cancer.
* Unstable liver disease (as defined by presence of ascites, encephalopathy, coagulopathy, esophageal or gastric varices, or persistent jaundice), cirrhosis, and/or known biliary abnormalities.
* Poorly controlled hypertension defined as ≥160 mmHg systolic or ≥100 mmHg diastolic measurements taken within 30 days prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of ENG or its formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Current use of drugs known to be contraindicated with ENG (see A5392 Prohibited and Precautionary Medications document on the PSWP).
* Use of any drugs known to: 1) induce CYP3A4 system within 30 days prior to study entry or 2) inhibit the CYP3A4 system within 1 week immediately prior to study entry (see A5392 Prohibited and Precautionary Medications document on the PSWP).
* Plans to use prohibited medications during the study (see A5392 Prohibited and Precautionary Medications document on the PSWP).
* For Group B study candidates only, prior use of LA CAB or RPV.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 14 days prior to study entry.
* Undiagnosed abnormal genital bleeding within 30 days prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-08-02 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
ENG PK parameter Area under the concentration-time curve (AUC0-24weeks) based on ENG PK samples obtained from individual participants | PK samples at pre-insertion, and 1, 4, 12 and 24 weeks post implant insertion
  AUC for each participant will be calculated from all available ENG concentrations measured over 24 weeks using the linear interpolation version of trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule uses linear interpolation between untransformed data up through Clast. Assay lower limit of quantification (LLoQ) for ENG is 0.025 ng/mL; values < LLoQ were imputed as 0 (if pre-dose) or as ½ the LLoQ, 0.0125 ng/mL (if post-dose).

SECONDARY OUTCOMES:
ENG PK parameter Area under the concentration-time curve (AUC0-12weeks) based on ENG PK samples obtained from individual participants | PK samples at pre-insertion, and 1, 4, and 12 weeks post implant insertion
  AUC for each participant will be calculated from all available ENG concentrations measured over 12 weeks using the linear interpolation version of trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule uses linear interpolation between untransformed data up through Clast. Assay lower limit of quantification (LLoQ) for ENG was 0.025 ng/mL; values < LLoQ were imputed as 0 (if pre-dose) or as ½ the LLoQ, 0.0125 ng/mL (if post-dose).
Probability of having ENG implant removed due to intolerance before 48 weeks | From insertion of implant to 48 weeks
  Probability estimated by method of Kaplan and Meier that censors when ENG implant removed for reasons other than intolerance
ENG PK parameter Area under the concentration-time curve (AUC0-48weeks) based on ENG PK samples obtained from individual participants | PK samples at pre-insertion, and 1, 4, 12, 24, 36 and 48 weeks post implant insertion
  AUC for each participant will be calculated from all available ENG concentrations measured over 48 weeks using the linear interpolation version of trapezoidal rule (i.e., noncompartmental technique) using the software package Phoenix WinNonLin (Certara®). This version of the trapezoidal rule uses linear interpolation between untransformed data up through Clast. Assay lower limit of quantification (LLoQ) for ENG was 0.025 ng/mL; values < LLoQ were imputed as 0 (if pre-dose) or as ½ the LLoQ, 0.0125 ng/mL (if post-dose).
ENG total concentration in serum | PK samples at pre-insertion, and 1, 4, 12, 24, 36 and 48 weeks post implant insertion
  ENG concentrations in ng/mL measured over 48 weeks. Assay lower limit of quantification (LLoQ) for ENG was 0.025 ng/mL; values < LLoQ were imputed as ½ the LLoQ, 0.0125 ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Weinberg, MD, Study Chair — University of Colorado Hospital CRS

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the AIDS Clinical Trials Group by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the AIDS Clinical Trials Group.
  * For what types of analyses? To achieve aims in the proposal approved by the AIDS Clinical Trials Group.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the AIDS Clinical Trials Group "Data Request" form at: https://actgnetwork.org/about-actg/templates-and-forms. Researchers of approved proposals will need to sign an AIDS Clinical Trials Group Data Use Agreement before receiving the data.

REFERENCES:
- See also: Related Info — http://www.actgnetwork.org